CLINICAL TRIAL: NCT00467441
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Investigate the Efficacy and Safety of VSF-173 and Matching Placebo in Healthy Male and Female Subjects With Induced Excessive Sleepiness
Brief Title: VSF-173 Study in Healthy Adult Volunteers for Treatment of Induced Excessive Sleepiness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VP-VSF-173-2001
Record Dates: First submitted 2007-04-26; First posted 2007-04-30 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-10

CONDITIONS: Excessive Somnolence

INTERVENTIONS:
Drug: VSF-173

SUMMARY:
The purpose of this study is to determine the safety and efficacy of VSF-173 compared to placebo in treatment of induced excessive sleepiness.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with no medical, psychiatric, or current sleep disorders
* Subject must sign a written consent form

Exclusion Criteria:

* Evidence of excessive daytime sleepiness
* History of sleep disorders
* Psychiatric or neurological disorders

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)

PRIMARY OUTCOMES:
Ability to stay awake as assessed by Maintenance of Wakefulness Test (MWT)

SECONDARY OUTCOMES:
Mood
Psychomotor performance
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Gunther Birznieks, Study Director — Vanda Pharmaceuticals
Locations (1):
- Vanda Investigational Site, Dijon, France